CLINICAL TRIAL: NCT05269745
Title: Influence of Immobilisation, Stretching and Activity on Morphological and Mechanical Properties of Spastic Muscle
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 25940
Record Dates: First submitted 2022-02-14; First posted 2022-03-08 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy, Spastic
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise; G2 Phase Cell Cycle Checkpoints

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immobilization group (IG) (Active Comparator): One group - immobilization group (IG) - will receive the standard treatment.
  Interventions: Other: Stretching through immobilisation (IG)
- Immobilization/Activity Group (IAG) (Experimental): The other group - Immobilization/Activity Group (IAG) - will be treated with a new approach.
  Interventions: Other: Stretching through immobilisation and activity (IAG)
- Control Phase (Other): Before the intervention with the orthotic treatment starts, a control phase of 8 weeks is planned.
  Interventions: Other: Control Phase

INTERVENTIONS:
Other: Stretching through immobilisation (IG) — The immobilization group (IG) will receive the standard treatment, a dynamic ankle-foot orthosis (AFO) for night and day use (23 hours per day)
  Other Names: IG
  Arms: Immobilization group (IG)
Other: Stretching through immobilisation and activity (IAG) — The Immobilization/Activity Group (IAG) will be treated with the same type of ankle-foot orthosis at night (8 hours) and for 6 hours during the day (altogether orthosis treatment 14 hours per day). The rest of the day (10 hours) children and adolescents will be using only the foot shell of orthoses (FS) without the lower leg shell, to secure the correct position of the foot and to allow a free motion at ankle joint with a good correction of the foot deformity (e.g. Pes equinovarus / equinovalgus, midfoot-break).
  Other Names: IAG
  Arms: Immobilization/Activity Group (IAG)
Other: Control Phase — Before the intervention with the orthotic treatment starts, a control phase of 8 weeks is planned. During this time, the individual orthoses for each subject are manufactured.
  Arms: Control Phase

SUMMARY:
Neurologic changes caused by cerebral palsy (CP) result in adaptation of muscle architecture and function (e.g. shortened muscles and contractures). Stretching through immobilization (orthotic treatment) is one of the common interventions to bring the spastic muscle to growth. Positive outcomes of stretching through immobilization are increased range of motion and improved function. On the other hand, immobilization leads to disuse muscle atrophy. Hence, we hypothesize that combining a stretching through immobilization and muscle activity while controlling for foot deformity could be a superior treatment approach, which should lead to improved muscle morphology as well as function. The aim of the study is to examine the influence of two orthotic treatments (a standard regime and one new approach) on spastic plantar flexor muscles in children and adolescents with CP. The standard regime (stretching through immobilisation) includes a dynamic AFO (ankle-foot orthosis) used during day and night. The new approach combines stretching through immobilisation and allows for plantarflexor activity due to an innovative construction of the orthotic device.

This prospective randomized controlled study will recruit 20 ambulant children and adolescents (aged 5 to 15 years) with cerebral palsy and equinus deformity (GMFCS = Gross Motor Function Classification System level I to III). Each child will be randomized and stratified according to age and GMFCS to one of two groups. The first group receives the standard treatment (stretching through immobilization) using custom-made ankle foot orthosis for 23 hours per day. The other group will be treated with the same orthosis at night (8 hours) and for 6 hours during the day but the remaining 10 hours will be treated with the foot shell only that corrects subtalar and Chopart joints but does not block the ankle joint movement, so that more activity of plantarflexors will be possible during the day. The intervention will last for 12 weeks. Each child will be examined at four occasions (8 weeks before intervention = control phase, at the beginning of the intervention and then 8 and 12 weeks later). The main outcome measure is the fascicle length measured using a 3D ultrasound (3DUS) imaging technique. Further parameters of interest span across the whole levels of ICF including clinical examinations, biomechanics of gait, muscle morphologic and mechanic properties and participations questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory children with spastic CP.
* Ability to accept and follow verbal instruction.
* Limited range of motion in ankle joint - maximal dorsiflexion with knee extended ≤ 5°
* Gross Motor Functional Classification System level I-III.
* Age 5-15 years.
* Willingness to participate.

Exclusion Criteria:

* Other than spastic form of CP (ataxic, athetoid or dystonic).
* Severe mental retardation.
* Normal range of motion in ankle joint
* Oral antispastic or muscle relaxing medication.
* History of orthopaedic surgery in the last 12 months.
* History of botulinum toxin type A application in the last six months.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in mechano-morphological muscle-tendon properties - muscle volume | Time Frame: baseline (T1), PRE-measurement (T2, 8 weeks), POST-measurement (T3, 16 weeks), FOLLOW-UP measurement (T4, 20 weeks)
  Gastrocnemius medialis muscle volume
Change in mechano-morphological muscle-tendon properties - fascile length | Time Frame: baseline (T1), PRE-measurement (T2, 8 weeks), POST-measurement (T3, 16 weeks), FOLLOW-UP measurement (T4, 20 weeks)
  Gastrocnemius medialis fascile length
Change in mechano-morphological muscle-tendon properties - unit length | Time Frame: baseline (T1), PRE-measurement (T2, 8 weeks), POST-measurement (T3, 16 weeks), FOLLOW-UP measurement (T4, 20 weeks)
  Gastrocnemius medialis muscle belly, tendon and muscle-tendon unit length
Change in mechano-morphological muscle-tendon properties - elongation | Time Frame: baseline (T1), PRE-measurement (T2, 8 weeks), POST-measurement (T3, 16 weeks), FOLLOW-UP measurement (T4, 20 weeks)
  Passive gastrocnemius medialis muscle belly, tendon and muscle-tendon unit elongation due to externally applied torque to the ankle joint [elongation in mm]
Change in mechano-morphological muscle-tendon properties - stiffness | Time Frame: baseline (T1), PRE-measurement (T2, 8 weeks), POST-measurement (T3, 16 weeks), FOLLOW-UP measurement (T4, 20 weeks)
  Passive gastrocnemius medialis muscle belly, tendon and muscle-tendon unit stiffness due to externally applied torque to the ankle joint [stiffness in N/mm]
Change in joint range of motion | Time Frame: baseline (T1), PRE-measurement (T2, 8 weeks), POST-measurement (T3, 16 weeks), FOLLOW-UP measurement (T4, 20 weeks)
  Ankle joint range of motion (maximal plantarflexion - maximal dorsiflexion)
Change in maximal isometric muscle strength | Time Frame: baseline (T1), PRE-measurement (T2, 8 weeks), POST-measurement (T3, 16 weeks), FOLLOW-UP measurement (T4, 20 weeks)
  Maximal isometric torque production (isokinetic dynamometry)
Change in gait characteristics | Time Frame: baseline (T1), PRE-measurement (T2, 8 weeks), POST-measurement (T3, 16 weeks), FOLLOW-UP measurement (T4, 20 weeks)
  Gait kinematics (joint angles [°]) and kinetics (joint moments [Nm/kg]) of the hip, knee, and ankle joints (3D motion capture). Joint angles [°] and moments [Nm/kg] will be combined to report changes in gait pattern.

SECONDARY OUTCOMES:
Change in self-reported gait, mobility, and functional performance - GOAL | Time Frame: baseline (T1), PRE-measurement (T2, 8 weeks), POST-measurement (T3, 16 weeks), FOLLOW-UP measurement (T4, 20 weeks)
  Gait Outcomes Assessment List (GOAL) Questionnaire
Change in self-reported gait, mobility, and functional performance - PODCI | Time Frame: baseline (T1), PRE-measurement (T2, 8 weeks), POST-measurement (T3, 16 weeks), FOLLOW-UP measurement (T4, 20 weeks)
  Pediatrics Outcomes Data Collection Instrument (PODCI) Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Habersack, BSc MSc, Principal Investigator — Medical University of Graz; Martin Svehlik, MD PhD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No
It is yet not decided if individual data will be shared with other researchers.